CLINICAL TRIAL: NCT01521273
Title: A Multiple Meal Study to Evaluate the Role of Phytic Acid From Beans on Human Iron Absorption
Brief Title: Iron Absorption From Biofortified Beans With Different Levels of Phytic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Rwa3
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Enrichment of Blood
Keywords: beans; biofortification; phytic acid; iron; iron isotopes; different phytic acid concentrations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- high iron bean with native phytic acid concentration (Experimental)
  Interventions: Other: Bean varieties
- normal iron bean with native phytic acid concentration (Experimental)
  Interventions: Other: Bean varieties
- high iron bean partially dephytinized (Experimental)
  Interventions: Other: Bean varieties
- normal iron bean partially dephytinized (Experimental)
  Interventions: Other: Bean varieties
- high iron bean totally dephytinized (Experimental)
  Interventions: Other: Bean varieties
- normal iron bean totally dephytinized (Experimental)
  Interventions: Other: Bean varieties

INTERVENTIONS:
Other: Bean varieties — 10 x 50 g/ arm

SUMMARY:
Iron deficiency and iron deficiency anemia are among the major health problems in the developing world. Women of childbearing age as well as children are the most vulnerable population groups. In Rwanda, more than 40% of the population is estimated to be anemic. A promising approach to combat iron deficiency in Rwanda is biofortification of beans. The average consumption of beans is about 150 g per person per day in Rwanda and beans are a major staple food. Traditional plant breeding has increased the iron content of certain bean varieties from about 5 to 11 mg/100g. Iron absorption from beans however is with about 2-3% low because of high phytate and high polyphenol contents. A recently conducted study in Rwanda showed that the total amount of iron absorbed from a biofortified high iron bean was similar to the amount of iron absorbed from a control bean, which had a 50% lower iron concentration. This was surprising since the subjects had a low iron status and where therefore expected to maximize iron absorption. However, it was concluded that the additional iron bred into the bean was not bioavailable most likely due to the strong inhibitory nature of phytate in the high iron bean. To clarify that, a multiple meal study (iron absorption study) in collaboration of the Human Nutrition Laboratory of ETH Zurich and the Medical Faculty of the National University of Rwanda is planned. Subjects will receive two different bean varieties (normal iron vs. high iron) in combination with other food ingredients typical for that region. The bean varieties will be served with native phytate concentration, partially dephytinized (50%) or totally dephytinized.

Subjects will be apparently healthy females of reproductive age (18-30y). Iron absorption will be determined by stable isotope techniques.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating women
* Between 18 and 40 years
* Below 65kg

Exclusion Criteria:

* Metabolic, chronic and gastro-intestinal disease
* Long-term medication
* Blood donation within 6 month before the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The impact of different bean phytic acid concentrations on iron absorption measured by stable iron isotope techniques | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, Prof. Dr., Study Director — Swiss Federal Institute of Technology
Locations (1):
- National University of Rwanda (NUR), Butare, Rwanda

REFERENCES:
- [Derived] Petry N, Egli I, Gahutu JB, Tugirimana PL, Boy E, Hurrell R. Phytic acid concentration influences iron bioavailability from biofortified beans in Rwandese women with low iron status. J Nutr. 2014 Nov;144(11):1681-7. doi: 10.3945/jn.114.192989. Epub 2014 Sep 3. PMID 25332466